CLINICAL TRIAL: NCT02125617
Title: uPAR in Blood From Zytiga® (Abiraterone) Treated Patients With Castration Resistant Prostate Cancer - a Predictive Marker of Response?
Brief Title: Urokinase Plasminogen Activator Receptor in Abiraterone Treated Patients With Castration Resistant Prostate Cancer
Acronym: uPARCRPC
Status: Terminated | Type: Observational
Why Stopped: Poor recruition
Sponsor: Kristoffer Rohrberg (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kristoffer Rohrberg, MD, Phd, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: uPARCRPC
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2015-11

CONDITIONS: Prostatic Neoplasms
Keywords: Castration-resistant prostate cancer; Abiraterone; Biomarker; Urokinase Plasminogen Activator Receptor; Plasma; Predictive markers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; Prednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Castration-resistant prostate cancer, Progression after taxane: Treated with abiraterone 1000 mg/day Prednisolone 10 mg/day
  Interventions: Drug: Abiraterone; Drug: Prednisolone

INTERVENTIONS:
Drug: Abiraterone — 1000 mg/day
  Other Names: Zytiga®
Drug: Prednisolone — 10 mg/day

SUMMARY:
The purpose of this study is to investigate cleavage products of the urokinase plasminogenactivator receptor (uPAR) in plasma from patients with castration resistant prostate cancer as a predictive marker of response to abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥18 years and male
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Received at least one but not more than two cytotoxic chemotherapy regimens for metastatic CRPC. At least one regimen must have contained a taxane such as docetaxel.
* Prostate cancer progression as assessed by the investigator with one of the following:

  * PSA progression according to Prostate Cancer Working Group 2 (PCWG2) criteria
  * Solid Tumors (RECIST) criteria or bone scans with or without PSA progression.
  * Radiographic progression in soft tissue according to Response Evaluation Criteria in
* Ongoing androgen deprivation with serum testosterone <2.0 nM
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Platelet count ≥100,000/μL
* Serum albumin ≥30 g/dL
* Serum creatinine <1.5 x upper limit of normal (ULN) or a calculated creatinine clearance ≥ 60 mL/min
* Serum potassium ≥3.5 mmol/L

Exclusion Criteria:

* Received abiraterone or MDV3100 in the past.
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection.
* Abnormal liver functions consisting of any of the following:

  * Serum bilirubin ≥1.5 x ULN (except for subjects with documented Gilbert's disease, for whom the upper limit of serum bilirubin is 51 µmol/l)
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.5 x ULN
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥95 mmHg); subjects with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy.
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or left ventricular ejection fraction (LVEF) of <50% at baseline.
* Known brain metastasis
* History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study drug
* Any acute toxicities due to prior chemotherapy or radiotherapy that have not resolved to a NCI-CTCAE (Version 4.0) Grade of ≤1. Chemotherapy induced alopecia and Grade 2 peripheral neuropathy is allowed.
* Use of other anticancer therapy including cytotoxic, radionucleotide, and immunotherapy; diethylstilbestrol; PC-SPES; spironolactone (ie, ALDACTONE, SPIRONOL); and other preparations such as saw palmetto thought to have endocrine effects on prostate cancer, within 4 weeks of Cycle 1 Day 1
* Prior systemic treatment with an azole drug (eg, fluconazole, itraconazole, ketoconazole) within 4 weeks of Cycle 1 Day 1
* Current enrolment in an investigational drug or device study or participation in such a study within 30 days of Day 1
* Condition or situation which, in the investigator's opinion, may put the subjects at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for this study include patients with CRPC in progression after therapy with a taxane who are candidates for therapy with standard second line therapy abiraterone.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2016-07-15 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Impact of baseline uPAR cleavage products on response. | 6 months
  Impact of baseline plasma concentration of uPAR cleavage products on overall response rate (ORR) defined as the proportion of patients with radiologic response according to the RECIST criteria or PSA-response.

SECONDARY OUTCOMES:
Impact of baseline plasma concentration of uPAR cleavage products on overall survival (OS). | 6 months
  Impact of baseline plasma concentration of uPAR cleavage products on overall survival (OS).
Impact of baseline plasma concentration of uPAR cleavage products on progression free survival (PFS). | 6 months
  Impact of baseline plasma concentration of uPAR cleavage products on progression free survival (PFS).
Impact of baseline plasma concentration of uPAR cleavage products on pain relief rate. | 6 months
  Impact of baseline plasma concentration of uPAR cleavage products on pain relief rate.
Impact of baseline plasma concentration of uPAR cleavage products on disease control rate (DCR). | 6 months
  Impact of baseline plasma concentration of uPAR cleavage products on disease control rate (DCR).
Impact of baseline plasma concentration of uPAR cleavage products on serious adverse events (SAE). | 6 months
  Impact of baseline plasma concentration of uPAR cleavage products on serious adverse events (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer S Rohrberg, MD, Phd, Study Chair — Rigshospitalet, Denmark
Locations (1):
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark